CLINICAL TRIAL: NCT03597815
Title: Examining the Relationship Between Diabetic Macular Edema and Obstructive Sleep Apnea: Prevalence, Association and Impact.
Brief Title: Diabetic Macular Edema - Obstructive Sleep Apnea Relationship Study
Acronym: DME-OSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: DME-OSA
Record Dates: First submitted 2018-07-03; First posted 2018-07-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Macular Edema; Sleep Apnea; Non Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — aflibercept

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DME positive, OSA positive: Visit 1: Baseline DME Treatment. Includes first EYELEA(aflibercept) injection. (DME positive patients will receive a minimum of 6 injections with the first five occurring at 1-month intervals and the sixth occurring two months after the fifth. Further injections will be provided at the discretion of the ophthalmologist in according to the treat and extend protocol of Eylea to ensure the DME is resolved by the end of the study.) Each injection is 2 mg (0.05 mL). Visit 2: Diagnosis of OSA - Overnight sleep study Visit 3: 1 month follow up post-CPAP initiation Visit 4: 6-month visit post DME initial treatment Visit 5: 2-3 month follow up - titration study (at sleep lab) Visit 6: 12-month visit post DME initial treatment in the OSA- group and at least 3 months post CPAP initiation in the OSA+ group Visit 7: 12-month sleep apnea follow up
  Interventions: Drug: Aflibercept 40 MG/ML [Eylea]; Diagnostic Test: OSA diagnostic test - overnight sleep study; Device: CPAP therapy for OSA positive patients
- DME positive, OSA negative: Visit 1: Baseline DME Treatment Includes first EYELEA(aflibercept) injection. (DME positive patients will receive a minimum of 6 injections with the first five occurring at 1-month intervals and the sixth occurring two months after the fifth. Further injections will be provided at the discretion of the ophthalmologist in according to the treat and extend protocol of Eylea to ensure the DME is resolved by the end of the study.) Each injections is 2 mg (0.05 mL). Visit 2: Diagnosis of OSA - Overnight sleep study Visit 3: 6-month visit post DME initial treatment Visit 4: 12-month visit post DME initial treatment in the OSA- group and at least 3 months post CPAP initiation in the OSA+ group
  Interventions: Drug: Aflibercept 40 MG/ML [Eylea]; Diagnostic Test: OSA diagnostic test - overnight sleep study
- DME negative (NPDR positive), OSA positive: no injections needed. Visit 1: Baseline NPDR diagnosis Sleep lab visits Visit 2: Diagnosis of OSA - Overnight sleep study Visit 3: 1 month follow up post-CPAP initiation Visit 4: 2-3 month follow up - titration study Visit 5: 12-month sleep apnea follow up
  Interventions: Diagnostic Test: OSA diagnostic test - overnight sleep study; Device: CPAP therapy for OSA positive patients
- DME negative (NPDR positive), OSA negative: no injections needed. Visit 1: Baseline NPDR diagnosis Visit 2: Diagnosis of OSA - Overnight sleep study
  Interventions: Diagnostic Test: OSA diagnostic test - overnight sleep study

INTERVENTIONS:
Drug: Aflibercept 40 MG/ML [Eylea] — Intravitreal injection, form of anti-VEGF therapy
  Groups: DME positive, OSA negative; DME positive, OSA positive
Diagnostic Test: OSA diagnostic test - overnight sleep study — Overnight with specialist care in hospital - heart, lung and brain activity monitored.
Device: CPAP therapy for OSA positive patients — positive airway pressure ventilator, applies mild air pressure in a continuous basis to keep the airways continuously open in patients who are able to breath spontaneously on their own.
  Groups: DME negative (NPDR positive), OSA positive; DME positive, OSA positive

SUMMARY:
The purpose of this study is to evaluate the relationship between DME and obstructive sleep apnea (OSA). OSA impacts millions of North Americans, many of whom are undiagnosed. The investigators aim to evaluate if a relationship exists between the two diseases, whether or not the severity of OSA impacts the severity of DME, and whether treating OSA results in better treatment outcomes for DME. The study will involve the standard of care provided for both DME (involving anti-VEGF injections) and OSA (involving continuous positive airway pressure [CPAP] machine).Approximately 150 subjects are expected to be enrolled in this study.

In summary:

Question 1: Is there a correlation between DME and OSA? Question 2: Is there a relationship between the severity of DME (CRT and vision) and OSA (AHI index)? Question 3: Does treating OSA result in improving DME metrics, and does it neutralize the outcomes at 1 year compared to OSA negatives.

DETAILED DESCRIPTION:
A 12 month, non-randomized, controlled, prospective study evaluating the relationship between diabetic macular edema (DME) and obstructive sleep apnea (OSA).

Subjects eligible for the inclusion in the study will be grouped based on their diagnosis: DME & OSA positive, DME positive only, OSA positive only, and DME & OSA negative. All DME positive patients (irrespective of OSA status) will receive the standard of care treatment with anti-VEGF using Eylea in a standardized treat and extend protocol.

All patients will undergo baseline ophthalmologic examinations as part of a regular clinic visit including best-corrected visual acuity, intraocular pressure, slit lamp exam, dilated retinal exam, fluorescein angiography and optical coherence tomography (OCT). Diagnosis of diabetic macular edema will be confirmed with standard domain OCT. Diagnosis of OSA will be confirmed through gold standard of overnight polysomnography.

During each visit, the intraocular pressure and perfusion of the optic nerve head will be monitored for patient safety.

DME positive patients will receive a minimum of 6 injections with the first five occurring at 1-month intervals and the sixth occurring two months after the fifth. Further injections will be provided at the discretion of the ophthalmologist in according to the treat and extend protocol of Eylea. Data for Visits 1 and 4 in Table 1 will be collected at the first and sixth injections whereas the other injection visits will be treated as regular office visits and not study visits.

The investigators aim to identify the presence of OSA using the gold standard testing of an overnight sleep study to determine the prevalence of OSA in the DME population. Further, the investigators will attempt to determine if there is a correlation of OSA by comparing it to non-DME patients who have NPDR.

The mechanism of OSA action on diabetic microvascular complications may involve increased inflammatory responses and oxidative stress pathways such as increased advanced glycation end products. By comparing the gold standard metric of severity index of OSA (Apnea-hypopnea index) to DME metrics (LogMAR Snellen vision and CRT) at the baseline of both disease diagnoses, the investigators can determine severity association.

The specific metrics of DME treatment (Vision, CRT, number of injections) will be compared to pre-CPAP data to determine what the impact of CPAP was (if any) on DME treatment metrics. Further, the investigators aim to compare the one-year post-CPAP DME treatment metrics against one-year non-CPAP/non-OSA patients to determine the relative impact against a control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Ability to understand and provide written consent
* Type II diabetes patients and evidence of Diabetic Retinopathy
* Patients with and without DME
* Able and willing to comply with all treatment and follow-up procedures

Exclusion Criteria:

* Contraindications to Eylea including: stroke within the past month, ocular or periocular infection, active intraocular inflammation, hypersensitivity to Eylea and/or its excipients.
* Contraindication to CPAP including: severe bullous lung disease, pneumothorax, pathologically low blood pressure, dehydration, cerebrospinal fluid leak, recent cranial surgery, or trauma
* Any other types of retinal diseases such as retinal detachment
* Any other types of macular disease such as age-related macular degeneration
* Mental capacity to comply is impaired (i.e. dementia)
* Pregnant or breastfeeding women
* Participation in any drug or device clinical investigation within 30 days prior to entry into the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Uptown Eye Clinic who comply with the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Presence of DME | First visit, 0 months
Presence of OSA | First visit, 0 months
Snellen visual acuity | 12 months
Apnea-Hypopnea Index | 12 months

SECONDARY OUTCOMES:
Central Retinal Thickness | 12 months
  for DME +ve patients
Number of injections | 7 months +
  for DME +ve patients
CPAP compliance | 12 months
  for OSA+ patients

CONTACTS AND LOCATIONS:
Overall Officials: Sohel Somani, Principal Investigator — Uptown Eye
Locations (1):
- Uptown Eye Speicialists, Brampton, Otario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster GD, Sanders MH, Millman R, Zammit G, Borradaile KE, Newman AB, Wadden TA, Kelley D, Wing RR, Sunyer FX, Darcey V, Kuna ST; Sleep AHEAD Research Group. Obstructive sleep apnea among obese patients with type 2 diabetes. Diabetes Care. 2009 Jun;32(6):1017-9. doi: 10.2337/dc08-1776. Epub 2009 Mar 11. PMID 19279303
- [Background] Resnick HE, Redline S, Shahar E, Gilpin A, Newman A, Walter R, Ewy GA, Howard BV, Punjabi NM; Sleep Heart Health Study. Diabetes and sleep disturbances: findings from the Sleep Heart Health Study. Diabetes Care. 2003 Mar;26(3):702-9. doi: 10.2337/diacare.26.3.702. PMID 12610025
- [Background] Sacramento JF, Ribeiro MJ, Rodrigues T, Guarino MP, Diogo LN, Seica R, Monteiro EC, Matafome P, Conde SV. Insulin resistance is associated with tissue-specific regulation of HIF-1alpha and HIF-2alpha during mild chronic intermittent hypoxia. Respir Physiol Neurobiol. 2016 Jul;228:30-8. doi: 10.1016/j.resp.2016.03.007. Epub 2016 Mar 15. PMID 26993367
- [Background] Reichmuth KJ, Austin D, Skatrud JB, Young T. Association of sleep apnea and type II diabetes: a population-based study. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1590-5. doi: 10.1164/rccm.200504-637OC. Epub 2005 Sep 28. PMID 16192452
- [Background] Shiba T, Sato Y, Takahashi M. Relationship between diabetic retinopathy and sleep-disordered breathing. Am J Ophthalmol. 2009 Jun;147(6):1017-21. doi: 10.1016/j.ajo.2008.12.027. Epub 2009 Mar 9. PMID 19268888
- [Background] West SD, Groves DC, Lipinski HJ, Nicoll DJ, Mason RH, Scanlon PH, Stradling JR. The prevalence of retinopathy in men with Type 2 diabetes and obstructive sleep apnoea. Diabet Med. 2010 Apr;27(4):423-30. doi: 10.1111/j.1464-5491.2010.02962.x. PMID 20536514
- [Background] Banerjee D, Leong WB, Arora T, Nolen M, Punamiya V, Grunstein R, Taheri S. The potential association between obstructive sleep apnea and diabetic retinopathy in severe obesity-the role of hypoxemia. PLoS One. 2013 Nov 18;8(11):e79521. doi: 10.1371/journal.pone.0079521. eCollection 2013. PMID 24260240
- [Background] Leong WB, Jadhakhan F, Taheri S, Chen YF, Adab P, Thomas GN. Effect of obstructive sleep apnoea on diabetic retinopathy and maculopathy: a systematic review and meta-analysis. Diabet Med. 2016 Feb;33(2):158-68. doi: 10.1111/dme.12817. Epub 2015 Jul 4. PMID 26031931
- [Background] Mason RH, West SD, Kiire CA, Groves DC, Lipinski HJ, Jaycock A, Chong VN, Stradling JR. High prevalence of sleep disordered breathing in patients with diabetic macular edema. Retina. 2012 Oct;32(9):1791-8. doi: 10.1097/IAE.0b013e318259568b. PMID 22714043
- [Background] Mason RH, Kiire CA, Groves DC, Lipinski HJ, Jaycock A, Winter BC, Smith L, Bolton A, Rahman NM, Swaminathan R, Chong VN, Stradling JR. Visual improvement following continuous positive airway pressure therapy in diabetic subjects with clinically significant macular oedema and obstructive sleep apnoea: proof of principle study. Respiration. 2012;84(4):275-82. doi: 10.1159/000334090. Epub 2011 Dec 20. PMID 22189259

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03597815/Prot_SAP_000.pdf